CLINICAL TRIAL: NCT03073460
Title: The Role of Fetal Ductus Arteriosus in Predicting Spontaneous Labour at Term
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit any participants
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-037
Record Dates: First submitted 2017-02-15; First posted 2017-03-08 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound examination (Other): Participants will undergo an ultrasound examination at 40 weeks gestation to assess the fetal ductus arteriosis.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — This exam is performed at 40 weeks gestation

SUMMARY:
The exact mechanism stimulating the parturition in humans is still relatively unknown. Prostaglandins, by mediating cervical ripening and early stimulation of myometrial contractions, are likely to play a major role in the parturition process. Much of the unique fetal circulation is facilitated by the ductus arteriosus. Patency of the ductus arteriosus in utero is primarily maintained via prostaglandins which are highly expressed by smooth muscle cells located in the media of the ductus arteriosus. The aim of the study is to prospectively observe fetal ultrasound changes related to the ductus arteriosus. The primary objective is to prospectively assess, whether any changes in the fetal ductus arteriosus parameters exist at 40 weeks' gestation. The secondary objective is to investigate whether there is an association between the ductus arteriosus parameters and the time to delivery interval at 40 weeks' gestation.

DETAILED DESCRIPTION:
The rationale is to assess whether physiological responses that occur around the time of delivery, in both the mother and the fetus (elevated prostaglandins level), can be quantified using ultrasound of the fetal ductus arteriosus.

Whether or not the DA plays an active physiological role in the initiation of parturition is still unknown. Since prostaglandins are physiologically highly expressed within the fetal ductus arteriosus and also linked to some critical steps throughout parturition, it is hypothesized that structural and doppler flow pattern variations of the ductus arteriosus exist in the period surrounding the birth. These changes might occur before or after the intrinsic rise of prostaglandins and could be quantified using prenatal ultrasound of the fetal DA.

Identifying new physiological based variables that can assist in predicting the onset of labour, as the one suggested in the current study, is thus of great importance and may provide invaluable information into the overall future care and decision making during pregnancy, especially around the time of delivery. It may assist in creating future recommendations for pregnant women and improved healthcare standards during the delivery process.

ELIGIBILITY:
Inclusion criteria:

* Low risk singleton pregnancy at 40 weeks gestation.

Exclusion criteria:

* Smoking
* Underlying cardiac or respiratory illness
* Fetal growth restriction
* Medicated gestational hypertension or evolving preeclampsia
* Gestational diabetes controlled with insulin or oral medications
* Use of steroids for lung maturation in the current pregnancy
* Known major congenital anomalies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women with a singleton pregnancy
Enrollment: 0 (Actual)
Dates: Start 2016-06-02 (Estimated); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Fetal ductus arteriosus changes | 40 weeks gestation
  To prospectively assess whether any changes in blood flow in the fetal ductus arteriosus exist at 40 weeks' gestation.

SECONDARY OUTCOMES:
Time to delivery | From 40 weeks gestation to delivery
  To investigate whether there is an association between the ductus arteriosus blood flow and the time to delivery interval at 40 weeks' gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No